CLINICAL TRIAL: NCT02216006
Title: High Fresh Gas Flow After Intubation - A Randomized Clinical Trial
Brief Title: High Fresh Gas Flow After Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Erland Ostberg, M.D., Region Västmanland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dnr 2012/335
Record Dates: First submitted 2014-08-01; First posted 2014-08-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Atelectasis
Keywords: Atelectasis; Fresh gas flow; Prevention; Oxygenation; Anaesthesia
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group, conventional ventilatory settings (Active Comparator): Handling of the airway during induction and intubation is performed in a conventional manner.
  Initial ventilatory settings are also done in a conventional manner.
  Interventions: Procedure: Control group, conventional ventilatory settings
- High fresh gas flow, high minute ventilation (Active Comparator): Handling of the airway during induction and intubation is performed in a conventional manner.
  Immediately after confirming a successful intubation the effect of preoxygenation is eliminated with an anti-preoxygenation maneuver.
  Interventions: Procedure: High fresh gas flow, high minute ventilation

INTERVENTIONS:
Procedure: Control group, conventional ventilatory settings — Handling of the airway during induction and intubation is performed in a conventional manner.
  Initial ventilatory settings are also done in a conventional manner. As soon as correct position of the endotracheal tube is confirmed, controlled ventilation is started with a tidal volume of 7 mL/kg ideal body weight, PEEP 6 or 8 cm H2O (8 if BMI >25) and a respiratory frequency of 10. The fresh gas flow is set to 1 Liter per minute with an oxygen mixture of 40%, aiming for an inspired FiO2 of 30-35%.
  Unless the patient´s SpO2 falls below 90%, the FiO2 remains unchanged throughout the procedure.
  Arms: Control group, conventional ventilatory settings
Procedure: High fresh gas flow, high minute ventilation — Handling of the airway during induction and intubation is performed in a conventional manner.
  Immediately after confirming a successful intubation, the effect of preoxygenation is eliminated with a fresh gas flow of 10 L/min of air, delivered with volume controlled ventilation consisting of tidal volumes of approximately 15 ml/kg ideal body weight, a positive expiratory pressure of 10 cm H20 and a respiratory frequency of 10. As soon as the end tidal O2 reaches 25%, the ventilator settings are adjusted to normal values (same as in the control group), i.e. tidal volume 7 mL/kg ideal body weight, PEEP 6 or 8 cm H2O (8 if BMI >25). The mixture of oxygen in the fresh gas is increased to 40% and the fresh gas flow is set to 1 Liter per minute, aiming for an inspired FiO2 of 30-35%.
  Unless the patient´s SpO2 falls below 90%, the FiO2 remains unchanged throughout the procedure.
  Arms: High fresh gas flow, high minute ventilation

SUMMARY:
Atelectasis is common during and after general anesthesia. Atelectasis develops early if preoxygenation with 100% oxygen is used and continuously used during induction until endotracheal intubation. The investigators hypothesize that a rapid anti-preoxygenation maneuver immediately after confirming a successful intubation, reduces the area of atelectasis as investigated by computed tomography compared to a standard procedure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients, American Society of Anesthesiology (ASA) I-II
* Patients scheduled for orthopaedic day case surgery in general anaesthesia

Exclusion Criteria:

* ASA class III or higher
* Body Mass Index (BMI) 30 or higher
* Arterial oxygen saturation (SpO2) <94% breathing air
* Chronic Obstructive Pulmonary Disease (COPD)
* Ischemic heart disease
* Haemoglobin <100g/L
* Known or anticipated difficult airway and/or intubation
* Active smokers and ex-smokers with a history of more than 6 pack years
* Need for interscalene or supraclavicular regional anaesthesia with risk of phrenic nerve paralysis

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Atelectasis | Within 1-2 hours, just before emergence from anesthesia
  The area of atelectasis in the lungs is assessed by computed tomography (CT) 10 mm above the dome of the right diaphragm and expressed in cm2 and as % of the total lung area in the particular scan.

SECONDARY OUTCOMES:
Arterial blood gases | Within 2-3 hours perioperatively

CONTACTS AND LOCATIONS:
Overall Officials: Mats Enlund, MD, PhD, Study Chair — Landstinget i Värmland
Locations (1):
- Landstinget Västmanland, Köping, Västmanland County, Sweden